CLINICAL TRIAL: NCT05694325
Title: Biologic Characterization of Patients With Immune Thrombocytopenia (ITP)
Brief Title: Biologic Characterization of Patients With ITP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: ITP1222
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological evaluation (Other): characterization of biological features of enrolled ITP patients
  Interventions: Other: peripheral blood and bone marrow withdrawal

INTERVENTIONS:
Other: peripheral blood and bone marrow withdrawal — samples evaluation

SUMMARY:
This is a no-profit, multicenter, biological, non-pharmacologic study aimed to characterize from a biological point of view previously untreated primary ITP patients. To this end, peripheral blood, fecal and bone marrow samples will be collected at baseline and at 30 days and 180 days after treatment initiation - for each line of therapy - and the results of the biological analysis performed at each time point will then be compared.

DETAILED DESCRIPTION:
This is a no-profit, multicenter, biological, non-pharmacologic study aimed to characterize from a biological point of view ITP patients. Patients with previously untreated primary ITP who need first-line therapy will be included in the study.

To this end, peripheral blood, fecal and bone marrow samples will be collected at baseline and at 30 days and 180 days after treatment initiation. The same assessments will be repeated in case of any potential new line of therapy.

The results of the biological analysis performed at each time point will then be compared, in order to seek changes related to the natural history of the disease, the therapy administered and the response achieved.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary ITP, in need for first line treatment according to 2019 ITP consensus2.
2. Previously untreated patients. Patients who have already started first-line therapy because of life-threatening bleeding are admitted to the study if samples are collected within 24 hours of starting treatment. In such cases, as first-line treatment steroids and platelet transfusions would be preferable over high-dose IVIg. Treatment received before the collection of samples will be carefully documented.
3. Age ≥ 18 years
4. Signed written informed consent according to ICH/EU/GCP and national local laws.

Exclusion Criteria:

1. Secondary ITP. Patients with ANA positivity without a diagnosis of SLE are admitted to the study. As far as patients with ITP and antiphospholipid antibodies positivity, those with triple positivity (anti-beta2glicoprotein antibodies, anti-cardiolipin antibodies, lupus anticoagulans positivity) are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
B-cell mediated disease incidence | at baseline
  evaluation of percentage of patients with a predominant B-cell mediated disease

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Lucchini, Principal Investigator — SC Ematologia ASUGI
Locations (5):
- Italy (5):
  - UOC ematologia AOU di Bologna, Bologna
  - Ematologia e centro trapianti ASL Piacenza, Piacenza
  - Ematologia Policlinico Universitario A.Gemelli, Roma
  - Sc Ematologia Ospedale S.G. Battista Molinette - Università Degli Studi Di Torino, Torino
  - SC Ematologia ASUGI, Trieste